CLINICAL TRIAL: NCT04279847
Title: A Phase 1, Open-Label, Safety and Tolerability Study of INCB057643 in Participants With Myelofibrosis and Other Advanced Myeloid Neoplasms
Brief Title: Safety and Tolerability Study of INCB057643 in Participants With Myelofibrosis and Other Advanced Myeloid Neoplasms
Acronym: LIMBER
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 57643-103; 2023-506145-38-00 (Registry Identifier: EU CT Number); 2020-003532-25 (EudraCT Number)
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Myelofibrosis; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm Overlap Syndrome; Myeloproliferative Neoplasm; Relapsed or Refractory Primary Myelofibrosis; Secondary Myelofibrosis (Post-Polycythemia Vera Myelofibrosis, Post-Essential Thrombocythemia Myelofibrosis); ET (Essential Thrombocythemia)
Keywords: Myelofibrosis; myelodysplastic syndrome; myelodysplastic/myeloproliferative neoplasm overlap syndrome; myeloproliferative neoplasm; BET protein inhibitor; relapsed primary myelofibrosis; refractory primary myelofibrosis; secondary myelofibrosis; post-polycythemia vera myelofibrosis; post-essential thrombocythemia myelofibrosis; LIMBER; ET (essential thrombocythemia)
MeSH Terms: conditions — Primary Myelofibrosis; Myelodysplastic Syndromes; Myeloproliferative Disorders; Recurrence; Thrombocythemia, Essential | interventions — INCB057643; ruxolitinib

STUDY DESIGN:
Intervention Model Description: monotherapy and ruxoltinib combination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 : INCB057643 Monotherapy (Experimental): INCB057643 dose escalation and dose expansion
  Interventions: Drug: INCB057643
- Part 2 : INCB057643 Combination with Ruxolitinib (Experimental): Combination arm in dose escalation and dose expansion
  Interventions: Drug: INCB057643; Drug: Ruxolitinib

INTERVENTIONS:
Drug: INCB057643 — INCB057643 dose escalation and dose expansion.
Drug: Ruxolitinib — Ruxolitinib will be administered twice a day using the dose described for each Cohort in the protocol for Part 2.
  Arms: Part 2 : INCB057643 Combination with Ruxolitinib

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary efficacy of INCB057643 as monotherapy or combination with ruxolitinib for participants with myelofibrosis (MF) and other myeloid neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older at the time of signing the informed consent.
* Part 1 Monotherapy: Participants with confirmed diagnosis of relapsed or refractory MF (primary, or post-PV and post-ET), MDS, MDS/MPN, or ET who have received at least 1 prior line of therapy; are either refractory, relapsed, or intolerant to the last therapy; and there is no available therapy that would provide clinical benefit in the opinion of the investigator.

  * a. MF with measurable disease (palpable spleen and symptoms) as defined in the protocol and risk category of intermediate 2 or high according to DIPSS. MF participants must have received a JAK inhibitor(s), such as ruxolitinib.
  * b. ET participants should have disease refractory to hydroxyurea as defined by the protocol.
* Part 2 Combination with ruxolitinib.

  * a. Primary MF or secondary MFs (post-PV MF and post-ET MF), histologically or cytologically confirmed, with measurable disease (palpable spleen and symptoms) as defined in the protocol, either currently receiving ruxolitinib with suboptimal response or JAKi-naive.
  * b. Suboptimal response is defined as currently being treated with ruxolitinib monotherapy at a stable dose for ≥ 8 weeks immediately preceding the first dose of study treatment. One dose reduction due to toxicities within 8 weeks prior to Study Day 1 is permitted.
  * c. JAKi-naive is defined as those participants that have no prior use of any JAK inhibitor, including ruxolitinib, and;
  * d. Part 2 dose escalation: Risk category of intermediate-2 or high according to DIPSS.
  * e. Part 2 dose expansion: Risk category of intermediate-1, intermediate-2, or high according to DIPSS.
  * f. Part 2 dose expansion participants with chronic MF are defined as participants with bone marrow myeloblast percentage < 5% (not applicable if dry tap or blast count deemed not reliable by the investigator) and blast count in peripheral blood < 1% at screening and who are currently receiving ruxolitinib and having a suboptimal response.

Note: Study treatment should be delayed if peripheral blood blast count at baseline is > 3%; treatment should only be started with medical monitor approval.

* g. Part 2 dose expansion participants with accelerated-phase MF are defined as having either a bone marrow myeloblast percentage ≥ 5% to < 20% or a myeloblast percentage ≥ 10% in peripheral blood on 2 occasions at least 2 weeks apart, AND are currently receiving ruxolitinib and have a suboptimal response.
* h. Part 2 dose expansion participants with JAKi-naive MF are eligible to receive ruxolitinib, with peripheral blood blast count of < 10% at the screening hematology assessment.

  * Must not be a candidate for potentially curative therapy, including hematopoietic stem cell transplantation.
  * ECOG performance status 0 to 2.
  * Life expectancy ≥ 24 weeks.
  * Willingness to avoid pregnancy or fathering children based on criteria.
* a. Men must agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through 90 days after the last dose of study treatment and must refrain from donating sperm during this period. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed.
* b. Women of childbearing potential must have a negative serum pregnancy test at screening and before the first dose on Day 1 and must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed.
* c. Women of nonchildbearing potential (ie, surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥ 12 months of amenorrhea without any other medical reasons such as treatment with anticancer agents) are eligible.

Exclusion Criteria:

* Prior receipt of a BET inhibitor.
* Receipt of anticancer medications or investigational drugs within the protocol-defined interval before the first dose of study treatment. For Part 2 JAKi-naive, prior use of a JAK inhibitor (including ruxolitinib) and no use of experimental drug therapy for MF or any other standard drug (except hydroxyurea) used for MF or another indication within 3 months of starting study drug. For participants with suboptimal response to ruxolitinib, ruxolitinib will continue at the participants' current ongoing doses, no ruxolitinib washout is needed.
* Participants with exclusionary laboratory values at screening defined as, including, but not limited to,

  * a. Platelets. Part 1 (monotherapy dose expansion, MF): < 75 × 109/L. Part 1 (monotherapy dose expansion, ET): < 450 × 109/L. Part 2 (combination dose escalation and expansion): < 75 × 109/L. Part 2 (combination dose expansion, JAKi-naïve MF): < 100 × 109/L.
  * b. Hemoglobin: Participants unwilling to receive red blood cell transfusion to treat low hemoglobin levels are excluded.
  * c. ANC < 0.75 × 109/L.
* inadequate renal, hepatic and coagulation functions as defined in the protocol.
* Concurrent anticancer therapy other than the therapies being tested in this study.
* Participants who have received allogeneic hematopoietic stem cell transplantation within 6 months of enrollment (unless approved by the medical monitor), or have active graft versus-host disease, or have received immunosuppressive therapy following allogeneic transplant within 2 weeks of the first dose of study treatment.
* Unless approved by the medical monitor, may not have received autologous hematopoietic stem-cell transplant within 3 months before the first dose of study treatment.
* Significant concurrent, uncontrolled medical condition, including but not limited to, significant GI disorder, history of or current clinically significant or uncontrolled cardiac disease, history or presence of an abnormal ECG that, in the investigator's opinion, is clinically meaningful, and history of bleeding disorder or at a high risk of bleeding.
* Active bacterial, fungal, parasitic, or viral infection that requires therapy.
* Current use of prohibited medication as described in the protocol, including the use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half lives (whichever is longer) before the first dose of study treatment.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to approximately 9 months
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug monotherapy and in combination with ruxolitinib.

SECONDARY OUTCOMES:
Spleen Volume Response | Week 24
  Defined as achieving a protocol defined reduction at Week 24 relative to baseline as measured by MRI or CT scan.
Duration of a Spleen Volume Response from baseline (MF only) | Up to approximately 9 months
  Defined as the interval between the first spleen volume response and the date of the first measurement that no longer achieves the protocol defined criteria.
Symptom Response Rate (MF or ET) | Week 24
  Defined as the proportion of participants who achieve a protocol defined reduction in Total Symptomatic Score (TSS) relative to baseline as measured by the MPN-symptom assessment form (SAF) TSS.
Anemia Response (MF only) | Up to approximately 9 months
  A hemoglobin increase of 1.5 g/dL relative to baseline for any "rolling" 12-week period during the study treatment period, if transfusion independent (TI) at baseline or Achieving TI for any "rolling" 12-week period during the study treatment period, if transfusion dependent (TD) at baseline.
Duration of Anemia Response (MF only) | Up to approximately 9 months
  The interval from the first onset of anemia response to the earliest date of loss of anemia response that persists for at least 4 weeks or death from any cause for the TI participants at baseline or duration of RBC-TI period for participants achieving RBC-TI for at least 12 consecutive weeks during the study treatment period for the TD participants at baseline.
Changes in hemoglobin value from baseline (MF only) | Up to approximately 9 months
  Defined as the mean change from baseline in the hemoglobin value over 12-week treatment periods.
Red Blood Cell (RBC) Transfusion Burden (MF only) | Up to approximately 9 months
  Defined as the average number of RBC units per participant-month through Weeks 12, 24, and 48.
Overall response (ET only) | Up to approximately 9 months
  Defined as proportion of participants with complete response or partial response and hematological improvement/response as per definition for ET.
Duration of platelet count reduction or White Blood Cell (WBC) count reduction (ET only) | Up to approximately 9 months
  Defined as platelet count reduction or WBC count reduction lasting ≥ 12 weeks.
Bone Marrow (BM) Blast Complete Remission (MF, myelodysplastic syndrome (MDS), and MDS/myeloproliferative neoplasm (MPN)) | Up to approximately 9 months
  Defined as BM blasts achieving the protocol defined criteria.
BM Blast Partial Remission (MF, MDS, and MDS/MPN) | Up to approximately 9 months
  Defined as BM blasts achieving the protocol defined criteria.
Peripheral Blast Complete Remission (MF, MDS, and MDS/MPN) | Up to approximately 9 months
  Defined as peripheral blasts achieving the protocol defined criteria.
Peripheral Blast Partial Remission (MF, MDS, and MDS/MPN) | Up to approximately 9 months
  Defined as peripheral blast achieving the protocol defined criteria.
Durable Blast Complete or Partial remission (MF, MDS, and MDS/MPN) | Up to approximately 9 months
  Defined as achieving the protocol defined criteria.

CONTACTS AND LOCATIONS:
Locations (48):
- United States (19):
  - University of Alabama At Birmingham, Birmingham, Alabama
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Emory University-Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of Nj, New Brunswick, New Jersey
  - Nyu Langone Health - Long Island Hospital, Mineola, New York
  - Nyu Langone Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Huntsman Cancer Institute At University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Canada (3):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Jewish General Hospital, Montreal, Quebec
  - St Paul'S Hospital, Vancouver
- China (4):
  - Peking Union Medical College Hospital, Beijing
  - Nanfang Hospital_Southern Medical University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine (Fahzu), Hangzhou
  - Henan Cancer Hostipal, Zhengzhou
- Helsinki University Central Hospital, Helsinki, Finland
- Italy (6):
  - Aou Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori, Meldola
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga Di Orbassano, Orbassano
  - Centro Ricerche Cliniche Di Verona, Verona
- Japan (6):
  - Fujita Health University Hospital, Aichi
  - Chiba University Hospital, Chiba
  - National Cancer Center Hospital East, Chiba
  - University of Yamanashi Hospital, Chūō
  - Kyushu University Hospital, Fukuoka
  - Kumamoto Shinto General Hospital, Kumamoto
- Spain (5):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca
- United Kingdom (4):
  - United Lincolnshire Hospitals, Boston
  - Lincoln County Hospital, Lincoln
  - The Christie Nhs Foundation Trust Uk, Manchester
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No
Access to patient level data is not available for this study

REFERENCES:
- See also: Related Info — https://www.incyteclinicaltrials.com/limber/
- See also: Safety and Tolerability Study of INCB057643 in Participants With Myelofibrosis and Other Advanced Myeloid Neoplasms (LIMBER) — https://www.incyteclinicaltrials.com/study/?id=INCB%2057643-103&SearchTerm=INCB%2057643-103&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=